CLINICAL TRIAL: NCT00560768
Title: Predictive Risk Stratification Through T Variability in ICD Patients Without Pacing Indications
Acronym: Prediction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: KOLB / Principal investigator, Klinikum Coburg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Prediction - ITAC06 Eu; ITAC06 Eu
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Sudden Cardiac Death
Keywords: Risk stratification method, negative predictive value, fast ventricular arrhythmias, ICD; The negative predictive value of the T amplitude variance as a method for risk stratification for patients with an increased risk for SCD.
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Ovatio VR 6250 or DR6550

INTERVENTIONS:
Device: Ovatio VR 6250 or DR6550 — The study requires the implantation of locally approved material:
  * A right ventricular defibrillation lead
  * In case of use of a dual chamber ICD a right atrial pacing lead
  * A single chamber or dual chamber ICD manufactured by SORIN Group. At begin of the study this will be OVATIO VR model 6250 and OVATIO DR model 6550. Any new devices of same type manufactured by SORIN Group which will become locally approved during the conduction of the trial can be used in the study.
  Holter recording will be performed with a market approved recording system allowing high resolution ECG recording compatible with the analysis software for TVar.

SUMMARY:
The aim of the study is to assess the negative predictive value of the T amplitude variance as a method for risk stratification for patients with an increased risk for SCD.

ELIGIBILITY:
Inclusion Criteria:

Patient has been prescribed the implantation of an SORIN GROUP OvatioTM DR 6550 / VR 6250 system according to relevant currently-approved guidelines

* CHF since > 3 months and
* LVEF < 35% and
* NYHA class II or III

OR

* Prior Myocardial infarction since more than 4 weeks and
* LVEF < 30%

Exclusion Criteria:

* Documented spontaneous sustained ventricular tachycardia
* Prior implant of any device for ventricular cardiac pacing
* Existing indication for permanent ventricular pacing
* Myocardial infarction within 4 weeks prior to enrollment
* Arrhythmogenic RV-Dysplasia
* Brugada syndrome
* Long QT syndrome
* Performed within 3 months prior to enrollment or scheduled (within 3 months) cardiac revascularization (interventional or surgical)
* Any indication for CRT accordingly to the relevant currently-approved ACC/AHA1 or ESC35 guidelines for the implantation of a CRT system.
* Excisting or planned administration of amiodarone - initiation of amiodarone therapy during the run of the study will lead to immediate exclusion of the patient
* Permanent chronic atrial fibrillation / flutter
* Patient is unable to attend the scheduled follow-up visits at the participating centre
* Patient is already included in another ongoing clinical study
* Patient is unable to understand the objectives of the study
* Patient refuses to cooperate
* Patient is unable or refuses to provide informed consent
* Patient is minor (less than 18-year old)
* Patient has life expectancy of less than 1 year
* Patient is pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
TAV score and number of tachyarrhythmic events. | The two phases M0 - M12 and M12 - M24 will be examined separately. For each 12 months period the TAV score at its beginning and tachyarrhythmic events in the following 12 months will be assessed. The NPV will be calculated for both phases.

SECONDARY OUTCOMES:
TAV change | 12 months of follow up

CONTACTS AND LOCATIONS:
Overall Officials: BRACHMANN Johannes, PhD, Principal Investigator — Klinikum Coburg
Locations (30):
- United States (7):
  - Helen Kelle Hospital, Sheffield, Alabama
  - Valley Regional Arrhytmia Center, Tarzana, California
  - Piedmont Hospital, Atlanta, Georgia
  - CMC - NorthEast, Charlotte, North Carolina
  - Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Stafford M. Smith - Scranton Heart Institute, Clarks Green, Pennsylvania
  - Easton Cardiology, Easton, Pennsylvania
- Canada (4):
  - Grey-Nuns Hospital, Edmonton
  - Hotel-Dieu du CHUM, Montreal
  - Laval UH, Ste Foy, Québec
  - St. Michael's Hospital, Toronto
- Germany (18):
  - Herz-und Diabeteszentrum NRW, Bad Oeynhausen
  - Praxis Westend, Berlin
  - Universitatsklinik Krankenanstalten Bergmannsheil, Bochum
  - Medizinische Universitatsklinik, Bonn
  - Klinikum, Coburg
  - Landkrankhenhaus Coburg, Coburg
  - Evangelisches Krankenhaus, Düsseldorf
  - Evangelisches Krankhenhaus Düsseldorf, Düsseldorf
  - Kardiocentrum, Frankfurt
  - Kardiocentrum Frankfurt, Klinik Rotes Kreuz, Frankfurt
  - Städt Klinikum Lüneburg, Lüneburg
  - Johannes Gutenberg-Universitat, Mainz
  - Universitatklinikum Mainz, Mainz
  - Bogenhausen Städt. Krankenhaus, München
  - Krankenhaus Reinbeck St Adolf-Stift, Reinbeck
  - ST. Adolf Stift; Medizinische Klinik, Reinbek
  - Universitätsklinikum Würzburg, Würzburg
  - Medizinische Klinik und Poliklinik I / kardiologie, Würzburg
- Universitario La Fe, Valencia, Spain